CLINICAL TRIAL: NCT04758949
Title: A Two-cohort, Phase 2 Study of FL-101 as Neoadjuvant Therapy in Patients With Surgically Resectable Non-Small Cell Lung Cancer
Brief Title: FL-101 in Surgically Resectable Non-Small Cell Lung Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Flame Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FL-101-2001
Record Dates: First submitted 2021-02-10; First posted 2021-02-17 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Surgically Resectable; NSCLC; Nivolumab; FL-101; Placebo
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Nivolumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Cohort 2 will be randomized. The investigator and participants will be masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- FL-101 Monotherapy (Experimental): 30 patients will receive FL-101 prior to surgery.
  Interventions: Drug: FL-101
- FL-101 + Nivolumab (Experimental): 30 patients will receive FL-101 and Nivolumab prior to surgery.
  Interventions: Drug: FL-101; Drug: Nivolumab
- Nivolumab + Placebo (Active Comparator): 30 patients will receive Nivolumab and placebo prior to surgery.
  Interventions: Drug: Nivolumab; Drug: Placebo

INTERVENTIONS:
Drug: FL-101 — 200 mg administered intravenously every 2 weeks prior to surgery.
  Arms: FL-101 + Nivolumab; FL-101 Monotherapy
Drug: Nivolumab — 240 mg administered intravenously every 2 weeks prior to surgery.
  Arms: FL-101 + Nivolumab; Nivolumab + Placebo
Drug: Placebo — 200 mg administered intravenously every 2 weeks prior to surgery.
  Arms: Nivolumab + Placebo

SUMMARY:
Phase 2 trial to study FL-101 alone or in combination with nivolumab in patients who have surgically resectable Non-Small Cell Lung Cancer.

DETAILED DESCRIPTION:
A 2-Cohort, Phase 2, multicenter, parallel-design trial that will study patients with surgically resectable, stages I-IIIA, non-small cell lung cancer (NSCLC) . The clinical study will focus on whether FL-101 has direct anti-tumor activity when given alone prior to surgery, and if FL-101 improves the anti-tumor response when given in combination with nivolumab prior to surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Previously untreated and pathologically confirmed, surgically resectable Stage IA3, IB, II, or IIIA NSCLC of squamous or non-squamous histology.
2. ≥1 radiologically measurable tumor >2cm in diameter.
3. Smoking history ≥10 pack years.
4. Available tissue block for analysis from a core needle biopsy(or similar sample)
5. High-sensitivity C-reactive protein (hsCRP) level ≥2 mg/L

Exclusion Criteria:

1. Any prior exposure to chemotherapy, radiotherapy or systemic anti-cancer therapy (e.g., monoclonal antibody therapy) for lung cancer.
2. Malignancies other than NSCLC within 2 years prior to Cycle 1, Day 1, with the exception of those with a negligible risk of metastasis or death and with expected curative outcome
3. Currently participating in, or has participated in, a trial of an investigational agent within 4 weeks prior to the first dose of study treatment or 5 half-lives, whichever is longer and with recovery of clinically significant toxicities from that therapy.
4. Tumors known to express driver mutations of the EGFR or ALK pathways.
5. Known severe hypersensitivity (Grade ≥3) to FL-101, its active substance, or any of its excipients
6. Known history of human immunodeficiency virus or active Hepatitis B or Hepatitis C infection

Additional Exclusion Criteria for Patients with Stage II and III Disease

1. Prior treatment with anti-PD-1, anti-CTLA-4, or anti-PD-L1 therapeutic antibody or pathway-targeting agents
2. Treatment with systemic immunosuppressive medications (including but not limited to prednisone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor [anti-TNF] agents) within 2 weeks prior to Cycle 1, Day 1
3. Known severe hypersensitivity (Grade ≥3) to nivolumab or chemotherapy agents or to any of their excipients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-08-25 (Actual); Primary Completion 2021-12-22 (Actual); Study Completion 2021-12-22 (Actual)

PRIMARY OUTCOMES:
Number of patients with treatment related adverse events as assessed by NCI CTCAE v.5.0 | From time of first dose to 3 months after surgery
  To evaluate the tolerability, incidence and severity of AEs and SAEs graded according to NCI CTCAE v5.0 of FL-101 as monotherapy and in combination with nivolumab.

SECONDARY OUTCOMES:
Number of patients with treatment efficacy as assessed by pathological response (percentage of residual tumor) by independent pathology review. | At time of surgery (around 6-8 weeks)
  Cohort 1: To evaluate the activity of FL-101 neoadjuvant monotherapy in patients with Stage IA3 or IB NSCLC
  Cohort 2: To evaluate the effect of FL-101 in combination with nivolumab compared to nivolumab plus placebo in neoadjuvant therapy in patients with Stage II-IIIA NSCLC
Major Pathologic Response | At time of surgery (around 6-8 weeks after first dose)
  To determine major pathologic response (MPR), defined as ≤10 percent viable tumor
Complete Pathologic Response | At time of surgery (around 6-8 weeks after first dose)
  To estimate complete pathologic response (CPR), defined as the absence of residual invasive cancer in resected lung specimens and lymph nodes
Objective Response Rate (ORR) | At time of surgery (around 6-8 weeks after first dose)
  To estimate objective response rate (ORR) by RECIST 1.1
MRD measurement by ctDNA | From time of first dose to 3 months after surgery
  To describe the time course of minimal residual disease (MRD) response by ctDNA and recurrence in correlation with clinical response

OTHER OUTCOMES:
Plasma Concentration of FL-101 | From time of first dose up to 3 months after surgery
  To evaluate the pharmacokinetics of FL-101 in patients with NSCLC
Plasma IL-1β/IL-6 levels | From time of first dose up to 3 months after surgery
  To evaluate the effect of FL-101 on pharmacodynamic biomarkers
Serum hsCRP | From enrollment up to 3 months after surgery
  To evaluate the effect of FL-101 on pharmacodynamic biomarkers
Prevalence and incidence of Anti-FL-101 antibodies | From time of first dose up to 3 months after surgery
  To evaluate possible immunogenicity of FL-101

CONTACTS AND LOCATIONS:
Overall Officials: Cassandra Choe-Juliak, MD, Study Director — Flame Biosciences